CLINICAL TRIAL: NCT03813420
Title: Sleep Quality Among Physiotherapy Students and Its Relation to Quality of Life and Physical Activity Level
Brief Title: Sleep Quality of Physiotherapy Students Quality of Life and Physical Activity Level
Acronym: SleepQuality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Habibe Serap Inal, Prof.Dr., Istinye University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ISU
Record Dates: First submitted 2018-12-31; First posted 2019-01-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Sleep Quality; Quality of Life; Physical Activity
Keywords: Sleep quality; Body mass index; Active life; Academic performance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy students (Other): 1. Pittsburgh Sleep Quality Index-PSQI:The sleep quality was evaluated through the Turkish version of the PSQI containing 19 self-rated questions searching the sleep quality during the previous month
  2. International Physical Activity Questionnaire-IPAQ: The physical activity of the participants was assessed through the Turkish version of the International Physical Activity Questionnaire -Short Form (IPAQ-SF), which includes 6 questions searching the frequency (days per week) and duration (hours) of walking, as well as the intensity of physical activity in the last seven days.
  3. Short Form-36-SF-36: The Turkish version of SF-36 was used to understand the health related quality-of -life (HRQOL) of the participants over the past four weeks in eight health concepts.
  Interventions: Behavioral: Pittsburgh Sleep Quality Index (PSQI); Behavioral: International Physical Activity Questionnaire (IPAQ); Behavioral: The Short Form 36 Health Survey (SF-36)

INTERVENTIONS:
Behavioral: Pittsburgh Sleep Quality Index (PSQI) — The sleep quality was evaluated through the Turkish version of the PSQI containing 19 self-rated questions searching the sleep quality during the previous month. It has seven components as subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction.
  Each component is scored from 0 to 3, and the Global Pittsburgh Quality of Sleep (PQS) score is the sum of the scores of the seven components that is between 0 and 21. The higher Global PQS scores indicate poor sleep quality and the cut off score for poor sleep is 5 and over.
  Other Names: IPAQ, SF-36 Quality of life
Behavioral: International Physical Activity Questionnaire (IPAQ) — The physical activity of the participants was assessed through the Turkish version of the International Physical Activity Questionnaire -Short Form (IPAQ-SF), which includes 6 questions searching the frequency (days per week) and duration (hours) of walking, as well as low, moderate and vigorous physical activity that they engaged in during the last seven days prior to survey. Vigorous physical activity, defined by the questionnaire, referred to intense exercise that resulted in very rapid breathing and an elevated heart rate (e.g. intense weight lifting, aerobics, running, and cycling). Moderate physical activity was defined as less intense exercise that slightly heightened breathing and heart rate (e.g. less exertive cycling, fast walking, and light weight lifting).
  Other Names: Pittsburgh Sleep Quality Index, SF-36
Behavioral: The Short Form 36 Health Survey (SF-36) — The Turkish version of SF-36 was used to understand the health related quality-of -life (HRQOL) of the participants over the past four weeks in eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. Additionally, the psychometric evaluation of the SF-36 generated two summary scores as the Mental Health Component Score and the Physical Health Component Score that the higher scores indicate better HRQOL.
  Other Names: IPAQ, Pittsburgh Sleep Quality Index

SUMMARY:
There is a high prevalence of poor sleep quality among university students studying in different areas such as medicine, nursing, art, science, social work etc. and in different countries. However, the studies done especially for physiotherapy students, and in Turkey, as well, are not many. Therefore, we aimed to search the sleep quality among physiotherapy students, and observe the association between the health related quality of life and physical activity level of the physiotherapy students.

The physiotherapy students were included. Their quality of sleep will be assessed by Pittsburgh Sleep Quality Index. The physical activity will be searched by International Physical Activity Questionnaire, and SF-36 will be used to assess quality of life. Data is going to analyzed statistically

DETAILED DESCRIPTION:
Therefore, recent studies are focusing on the sleep quality of university students in different countries, and reporting that medical students pharmacy students, nursing students are experiencing poor quality of sleep. However, to our knowledge, studies done on sleep quality of students and especially the physiotherapy students are not available in Turkey, yet.

Hence, since the university students are one of the high risk groups for developing poor sleep quality, we aimed to evaluate if the sleep quality of the physiotherapy students in both gender are associated with their quality of life and physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Being physiotherapy and rehabilitation students
* Being the age between 18-26 years old
* Being voluntary to participate to the study

Exclusion Criteria:

* Not having any systemic disease
* Any expressed psychological condition

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 3 months
  The sleep quality of the students will be evaluated by means of the Turkish version of the Pittsburgh Sleep Quality Index through face-to-face interview. This assessment will provide us information about the type and duration of their sleep as well as their sleep efficiency, if there are any sleep disturbances or if they are using any sleep medications or not. Additionally, this will provide us about if the sleep quality affects their daytime functions.

SECONDARY OUTCOMES:
Physical activity | 3 months
  The physical activity of the participants will assessed through the Turkish version of the International Physical Activity Questionnaire -Short Form. The frequency (days per week) and duration (hours) of walking, the intensity of their physical activity as if they are low, moderately and vigorously physical active or not will be searched. This covers the duration of the last seven days prior to survey.

OTHER OUTCOMES:
Health related quality-of -life | 3 months
  The Turkish version of SF-36 will used to understand the health related quality-of -life of the participants over the past four weeks. The eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions will be searched. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Ekin Aktay Karlik, MSc, Study Chair — Istanbul University
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manzar MD, Zannat W, Hussain ME, Pandi-Perumal SR, Bahammam AS, Barakat D, Ojike NI, Olaish A, Spence DW. Dimensionality of the Pittsburgh Sleep Quality Index in the collegiate young adults. Springerplus. 2016 Sep 13;5(1):1550. doi: 10.1186/s40064-016-3234-x. eCollection 2016. PMID 27652123
- [Result] Almojali AI, Almalki SA, Alothman AS, Masuadi EM, Alaqeel MK. The prevalence and association of stress with sleep quality among medical students. J Epidemiol Glob Health. 2017 Sep;7(3):169-174. doi: 10.1016/j.jegh.2017.04.005. Epub 2017 May 5. PMID 28756825
- [Result] Chang SP, Shih KS, Chi CP, Chang CM, Hwang KL, Chen YH. Association Between Exercise Participation and Quality of Sleep and Life Among University Students in Taiwan. Asia Pac J Public Health. 2016 May;28(4):356-67. doi: 10.1177/1010539516645160. Epub 2016 Apr 28. PMID 27130632
- [Result] Elagra MI, Rayyan MR, Alnemer OA, Alshehri MS, Alsaffar NS, Al-Habib RS, Almosajen ZA. Sleep quality among dental students and its association with academic performance. J Int Soc Prev Community Dent. 2016 Jul-Aug;6(4):296-301. doi: 10.4103/2231-0762.186788. PMID 27583216